CLINICAL TRIAL: NCT03178474
Title: Efficacy of JINLINGGUAN and TOFER Formula in Formula-fed Chinese Term Infants: A Controlled Trial
Brief Title: Efficacy of JINLINGGUAN and TOFER Formula in Formula-fed Chinese Term Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yu-ming Chen, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Yili_trial01
Record Dates: First submitted 2017-06-02; First posted 2017-06-07 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Infant Formula Intolerance; Well-being
Keywords: infant formula; Clinical trial; Chinese infant; body growth; gut microbiota; Stool characteristics
MeSH Terms: interventions — Milk, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Researchers involved in laboratory tests will be blinded to the group status
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Breast-Fed Group (Active Comparator): The infants will be fed with human breast milk by their mother
  Interventions: Other: Breast milk
- TOFER Formula Group (Experimental): TOFER Infant formula,TOFER®: Infants will be fed by using TOFER® infant formula (Phase I baby formula) from baseline (about 5-14 days) to 13 weeks of age.
  Interventions: Other: TOFER Infant formula,TOFER®
- JINLINGGUAN Formula Group (Experimental): JINLINGGUAN Infant formula,PRO-KIDO™ I-PROTECH®: Infants will be fed by using JINLINGGUAN (PRO-KIDO™ I-PROTECH®) infant formula (Phase I baby formula) from baseline (about 5-14 days) to 13 weeks of age.
  Interventions: Other: JINLINGGUAN Infant formula,PRO-KIDO™ I-PROTECH®

INTERVENTIONS:
Other: JINLINGGUAN Infant formula,PRO-KIDO™ I-PROTECH® — JINLINGGUAN Infant formula,PRO-KIDO™ I-PROTECH®: a type of Phase I infant formula for 0-6 month infants, with a trademark of PRO-KIDO™ I-PROTECH®. The formula contains both OPO structured lipid and α+β patented protein (patent number: ZL200810241156.3).It was produced by Inner Mongolia Yili Industrial Group Co.Ltd.,China
  Arms: JINLINGGUAN Formula Group
Other: TOFER Infant formula,TOFER® — TOFER Infant formula,TOFER®: a type of Phase I infant formula for 0-6 month infants, with a trademark of TOFER®. The formula was characterized by (1) Moderate digestible small-molecule protein; and (2) BID® complex probiotics. It was produced by Inner Mongolia Yili Industrial Group Co.Ltd.,China
  Arms: TOFER Formula Group
Other: Breast milk — Breast milk: Human breast milk, provided and fed by the corresponding infant's mother
  Arms: Breast-Fed Group

SUMMARY:
Objective：The present trial aimed to assess efficacy and safety of Jin Ling Guan and Tofer infant formula on body growth, intestinal tolerance, gut microbiota and fecal residual nutrients as compared to breast-milk in term Chinese infants.

Participants：189 healthy termed-infants with ages of 5-14 days at the enrollment.

Study Design: A multiple-center, quasi-randomized,open labeled, controlled trial. Random allocation between the two infant formula.

Arms, Groups, and Intervention: (1) Breast milk-fed group: fed with human breast milk; (2) JINLINGGUAN Formula Group：fed with JINLINGGUAN infant formula (PRO-KIDO™ I-PROTECH®, Phase I); (3) TOFER Formula Group: feeding TOFER infant formula (TOFER®, Phase I). Random allocation performed between the two formula groups.

Intervention Duration: 12 weeks.

Visits: 1 week(baseline), 7 and 13 weeks of age

Outcome measures: (1) General information, general health and wellbeing, regular body check;(2) Anthropometric parameters: body length, body weight, and head circumferences; (3) Stool characteristics (color , volume, stool consistency, and frequency;(4)Behavior and habits; (5) Gut microbiota; (6) Residual nutrients in feces (nitrogen,total fat, fatty acids, minerals); (7) adverse events and concomitant medications; (8) compliance. Slopes of changes from baseline to 6 and 12 weeks post intervention in anthropometric parameters, stool characteristic index, fecal residual nutrients, pattern score of gut microbiota, behavior and habit index were be calculated.

ELIGIBILITY:
Inclusion Criteria:

* The mother had unequivocally decided not to breast-feed (for formula fed infants) or to breastfeed (for human milk fed infants)
* Term infant of Chinese origin born at 37-42 gestation weeks
* Birth weight: 2500-4000g
* The infant is apparently healthy at birth and entry to study
* Apgar after 5 minutes >7
* age at the enrollment: 5-14 days

Exclusion Criteria:

* Mother health condition: (psychological or physical) or socioeconomic problems that may interfere with the mother's ability to take care of her infant
* The infant suffers from a major congenital abnormality or chromosomal disorder with a clinical significance that can be detected at birth
* The infant suffers/ed from a disease requiring mechanical ventilation or medication treatment at the first week after birth (not including photo treatment for infantile hepatitis)
* The infant suffers from any suspected or known metabolic or physical limitations interfering with feeding or normal metabolism

Ages: 5 Days to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2015-12-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-12-30 (Estimated)

PRIMARY OUTCOMES:
Average Change Rate of Stool Characteristic Index from Baseline to 6 and 12 weeks | 0, 6, 12 weeks
  Slope of change at 0, 6 and 12 weeks in Stool Characteristic Index: calculated using stool color (using sample pictures), volume (small, normal or large using sample picture scale), stool consistency (runny, mushy, soft, formed or hard), and frequency
Average Change Rate of Fecal Residual Nitrogen from Baseline to 6 and 12 weeks | 0, 6, 12 weeks
  Slope of change at 0, 6 and 12 weeks in Fecal Residual Nitrogen
Average Change Rate of Fecal Residual Fat from Baseline to 6 and 12 weeks | 0, 6, 12 weeks
  Slope of change at 0, 6 and 12 weeks in fecal residual total fat
Average Change Rate of Fecal Residual Calcium from Baseline to 6 and 12 weeks | 0, 6, 12 weeks
  Slope of change at 0, 6 and 12 weeks in fecal residual calcium

SECONDARY OUTCOMES:
Average Change Rate of an Index of General health and wellbeing from Baseline to 6 and 12 weeks | 0, 6, 12 weeks
  Slope of change at 0, 6 and 12 weeks in Index of General health and wellbeing, calculated from diseases (cold, diarrhea, bronchitis, pneumonia), doctor visits, gastro symptoms,etc.
Average Change Rate of Behavior and Habit Score from Baseline to 6 and 12 weeks | 0, 6, 12 weeks
  Slope of change at 0, 6 and 12 weeks in Behavior and Habit Score assessed by infant behavior questionnaires
Average Change Rate of body length from Baseline to 6 and 12 weeks | 0, 6, 12 weeks
  Slope of change at 0, 6 and 12 weeks in body length
Average Change Rate of Body Weight from Baseline to 6 and 12 weeks | 0, 6, 12 weeks
  Slope of change at 0, 6 and 12 weeks in body weight
Average Change Rate of Head Circumference from Baseline to 6 and 12 weeks | 0, 6, 12 weeks
  Slope of change at 0, 6 and 12 weeks in head circumference
Average Change Rate of Gut Microbiota Pattern Score from Baseline at 6 and 12 weeks | 0, 6, 12 weeks
  Slope of change at 0, 6 and 12 weeks in gut microbiota pattern score from 16S RNA sequencing
Average Change Rate of Pattern Score of Fecal Residual Fatty acids from Baseline at 6 and 12 weeks | 0, 6, 12 weeks
  Slope of change at 0, 6 and 12 weeks in the pattern score of fecal residual fatty acids

OTHER OUTCOMES:
Average Change Rate of Fecal Residual Iron from Baseline at 6 and 12 weeks | 0, 6, 12 weeks
  Slope of change at 0, 6 and 12 weeks in fecal residual iron
Average Change Rate of Fecal Residual Zinc from Baseline at 6 and 12 weeks | 0, 6, 12 weeks
  Slope of change at 0, 6 and 12 weeks in fecal residual zinc

CONTACTS AND LOCATIONS:
Overall Officials: Yuming Chen, Ph.D., Principal Investigator — Sun Yat-sen University
Locations (3):
- China (3):
  - Lankao Hospital, Kaifeng, Henan
  - Shaoyang Center Hospital, Shaoyang, Hunan
  - Nanxiong Hospital, Shaoguan

IPD SHARING:
Plan to Share IPD: No